CLINICAL TRIAL: NCT07256145
Title: Comparison Between the Efficacy of Ultrasound-guided Erector Spinae Plane Block and Conventional Treatment for Pain Management in Patients With Post-herpetic Neuralgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0307429
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Post-Herpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injection group (Experimental)
  Interventions: Procedure: erector spinae plane block
- conventional group (No Intervention)

INTERVENTIONS:
Procedure: erector spinae plane block — erector spinae plane block with steroids
  Arms: Injection group

SUMMARY:
The present study aims to evaluate the efficacy of ultrasound-guided erector spinae plane block with steroids to relieve pain in cases of post-herpetic neuralgia, patient satisfaction, and record any complications post-injection.

DETAILED DESCRIPTION:
The current study will be conducted as a single-blinded prospective randomized controlled study to evaluate the efficacy of ultrasound-guided erector spinae plane block with steroids to relieve pain in cases of post-herpetic neuralgia.

All patients will be evaluated by:

* Full history taking: including age, sex, presence of co-morbid conditions as well as the presenting complaint.
* Clinical examination and routine lab investigations that include:

  * Complete blood count (CBC).
  * Fasting blood glucose (FBG).
  * Coagulation profile (bleeding time, prothrombin time, prothrombin activity, international normalized ratio).

Measurements:

Patients will be followed up at 24 hours, 1 week, and 6 weeks after injection.

The following measurements will be recorded:

1. Pain will be assessed pre- and post-injection using VAS score at 24 hours, 1 week, and 6 weeks post-injection.
2. Need for analgesic intake post-injection will be assessed at the follow-up periods.
3. Patient satisfaction using the SAPS score.
4. Complications post-injection as pain, irritation or infection will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with post-herpetic neuralgia not responding to medical treatment.

Exclusion Criteria:

- 1- Patient refusal 2- Age less than 20 years or older than 70 years. 3- Systemic Infection. 4-Patients with dementia or other diseases that could have impaired their memory or cognitive function.

5- Immunocompromised patients, severe osteoporosis, and uncontrolled diabetes mellitus.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of ultrasound-guided erector spinae plane block with steroids to relieve pain in cases of post-herpetic neuralgia | 6 weeks
  by VAS score

SECONDARY OUTCOMES:
Patient satisfaction | 6 weeks
  SAPS score
Complications | 6 weeks
  As pain, irritation or infection

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Alexandria, Aleexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided